CLINICAL TRIAL: NCT03767205
Title: The Effect of a Ankle Assist Robot on Gait Function and Cardiopulmonary Metabolic Efficiency in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-06-128
Record Dates: First submitted 2018-12-02; First posted 2018-12-06 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2018-12

CONDITIONS: Stroke; Gait, Hemiplegic
Keywords: gait function; Metabolic energy expenditure; ankle assist robot
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stroke patients (Experimental): All participants perform overground walking and treadmill waking in three conditions (with robot-torque on/with robot-torque off/without robot).
  Interventions: Device: Ankle Assist Robot

INTERVENTIONS:
Device: Ankle Assist Robot — 1. overground walking in three conditions (with robot-torque on/with robot-torque off/without robot). During overground walking, gait function was measured using motion analysis, sEMG, and force plate
  2. treadmill waking in three conditions (with robot-torque on/with robot-torque off/without robot). During treadmill walking, the metabolic energy expenditure was measured using a portable cardiopulmonary metabolic system (Cosmed K4b², Rome, Italy).

SUMMARY:
The aim of this study was to identify the assistance effect of Ankle Assist Robot v1 developed by Samsung Advanced Institute of Technology (Samsung Electronics Co, Ltd., Korea) by comparing

1. gait function during overground gait in three conditions (with robot-assist torque on/with robot-assist torque off/without robot)
2. the energy expenditure during treadmill gait in three conditions (with robot-assist torque on/with robot-assist torque off/without robot)

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients with hemiplegia over 19 years old
* Ischemic or hemorrhagic stroke patients over 3 months of onset
* Functional Ambulation Category Scale with 3 or more scales

Exclusion Criteria:

* Stroke patients who have difficulty in walking independently regardless of assistive devices due to problems such as visual field defects or fractures
* Stroke patients with walking difficulty due to serious cognitive problems
* Patients with a foot size of 230 mm or less or a stroke of 280 mm or more that are not suitable for wearing ankle assist robot
* Stroke patients at risk of falling when walking with severe dizziness
* Modified ashworth scale (MAS) Stroke patients over 3
* Pregnant woman
* People with mental illness and psychiatric medication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change on gait speed in different three conditions | 20minutes
  All participants perform overground walking in different three conditions (with robot-torque on/with robot-torque off/without robot) to assess the change of gait speed using a motion analysis.

SECONDARY OUTCOMES:
Change on gait function in different three conditions (kinematic) | 20minutes
  All participants perform overground walking in different three conditions (with robot-torque on/with robot-torque off/without robot) to assess the change of kinematic using a motion analysis.
Change on gait function in different three conditions (kinetic) | 20minutes
  All participants perform overground walking in different three conditions (with robot-torque on/with robot-torque off/without robot) to assess the change of kinetic using a force plate.
Change on gait function in different three conditions (muscle activation) | 20minutes
  All participants perform overground walking in different three conditions (with robot-torque on/with robot-torque off/without robot) to assess the change of muscle activation using a surface EMG.
Change on metabolic energy expenditure in different three conditions | 1 hour
  All participants perform treadmill walking in different three conditions (with robot-torque on/with robot-torque off/without robot) to assess the change of metabolic energy expenditure using a portable cardiopulmonary metabolic system (Cosmed K4b², Rome, Italy).

CONTACTS AND LOCATIONS:
Overall Officials: YunHee Kim, Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee SH, Kim J, Lee HJ, Kim YH. A wearable ankle-assisted robot for improving gait function and pattern in stroke patients. J Neuroeng Rehabil. 2025 Apr 22;22(1):89. doi: 10.1186/s12984-025-01624-w. PMID 40264191